CLINICAL TRIAL: NCT04598425
Title: Cognitive Behavioral Therapy for Insomnia (CBTi) in Patients With Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Kåre Osnes, Principal Investigator, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00058 (PVO DS)
Record Dates: First submitted 2020-07-06; First posted 2020-10-22 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Insomnia; Insomnia Chronic; Insomnia Due to Mental Disorder; Insomnia, Psychophysiological; Sleep Disorder; Sleep Initiation and Maintenance Disorders; Sleep Disturbance; Mental Illness; Psychological Disorder; Depression, Anxiety
Keywords: Insomnia; Insomnia and co-morbid mental illness; Cognitive behavioral therapy for insomnia; CBTi
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Parasomnias; Mental Disorders; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive behavioral therapy for insomnia (CBTi) (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia (CBTi)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia (CBTi) — Patients will undergo a 7 sessions course in cognitive behavioral therapy for insomnia.

SUMMARY:
Insomnia is common in patients with co-morbid mental illness and sleeping difficulties is a frequent complaint in most psychological disorders. Mental illness may cause sleep problems, however, sleep problems like insomnia, may also cause or exacerbate mental illness. Insomnia may aggravate symptoms of depression, anxiety and fatigue, and reduce daily functioning in patients with co-morbid insomnia and mental illness. This project aims to evaluate a course offered to patients with insomnia and mental illness at Diakonhjemmet Hospital. The course is based on cognitive behavioral therapy, a documented treatment for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years with insomnia and co-morbid mental illness.
* Is a patient and receiving treatment for mental illness at Department of Psychiatry, Diakonhjemmet Hospital, at time of referral to the course

Exclusion Criteria:

* Unable to provide informed consent
* Unable to read and/or understand Norwegian
* Unable to complete a survey
* Severe mental disorder, e.g. schizophrenia and bipolar disorder type I
* Mental retardation or dementia
* Known substance abuse
* Other sleep disorder, e.g. narcolepsy and hypersomnia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in severity of insomnia | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Insomnia Severity Index (ISI; Minimum value = 0; Maximum value = 4. Higher scores mean worse outcome) to assess for any changes in symptoms of insomnia.
Change in symptoms of insomnia | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Bergen Insomnia Scale ( Minimum value = 0; Maximum value = 7. Higher scores mean worse outcome) to assess for any changes in symptoms of insomnia.

SECONDARY OUTCOMES:
Change in sleep efficiency | Calculations of sleep efficiency at baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course, will be compared.
  All patients included in the study will be asked to keep a sleep diary for the whole duration of the course. Sleep efficiency will be calculated based on the sleep diary.
Change in dysfunctional beliefs and attitudes about sleep | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Dysfunctional Beliefs and Attitudes about Sleep scale (DBAS-16; Minimum = 0; Maximum = 10. Higher values mean worse outcome) to assess for any changes in dysfunctional beliefs and attitudes about sleep.
Change in daytime rumination about tiredness and negative consequences of lack of sleep | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Daytime Insomnia Symptom Response Scale (DISRS; Minimum = 1; Maximum = 4. Higher values mean worse outcome) to assess for any changes in rumination about insomnia symptoms.
Change in compliance with sleep hygiene measures | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Sleep Hygiene Index (SHI-13; Minimum value = 1; Maximum value = 5. Higher values mean worse outcome) to assess for any changes in compliance with sleep hygiene measures.
Change in symptoms of depression | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Patient Health Questionnaire-9 (PHQ-9; Minimum value = 0; Maximum value = 3. Higher values mean worse outcome) to assess for any changes in symptoms of depression.
Change in symptoms of anxiety | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Generalized Anxiety Disorder Scale-7 (GAD-7; Minimum value = 0; Maximum value = 3. Higher values mean worse outcome) to assess for any changes in symptoms of anxiety.
Change in somatic symptoms | At baseline (before first session), at session 6 (last ordinary session, 5-7 weeks after baseline), at session 7 (2 months after last ordinary session) and 6 months after completing the course.
  All patients included in the study will be asked to complete the Somatic Symptom Scale-9 (SSS-8; Minimum value = 0; Maximum value = 4. Higher value mean worse outcome) to assess for any changes in somatic symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Kåre Osnes, M.D., Ph.D., Principal Investigator — Department of Psychiatry, Diakonhjemmet Hospital, Oslo, Norway
Locations (1):
- Department of Psychiatry, Diakonhjemmet Hospital, Oslo, Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No